CLINICAL TRIAL: NCT00677963
Title: Contrast-enhanced Ultrasound and Magnetic Resonance Imaging for the Evaluation of Neovascularisation in Carotid Artery Plaques
Brief Title: Contrast-enhanced Ultrasound (CE-US) and Magnetic Resonance Imaging (MRI): Evaluating Plaque Neovascularisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Werner H Mess/MD, PhD, Department of Clinical Neurophysiology, University Medical Center Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC 08-2-019
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Carotid Artery Stenosis; Atherosclerosis
Keywords: carotid; atherosclerosis; arteriosclerosis; plaque; neovascularization; carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis; Atherosclerosis; Arteriosclerosis; Plaque, Amyloid; Neovascularization, Pathologic | interventions — Sulfur Hexafluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Patients with symptomatic 70-99% carotid stenosis who are operated on.
  Interventions: Drug: sulphur hexafluoride, gadopentate dimeglumine

INTERVENTIONS:
Drug: sulphur hexafluoride, gadopentate dimeglumine — CE-US, using 2 x 2.4 ml sulphur hexafluoride and MRI, using 1 x 0.2 ml/kg gadopentate dimeglumine

SUMMARY:
The first goal of this study is to investigate whether CE-US is able to accurately identify and quantify neovascularisation in carotid artery plaques. Since this is one of the first studies systematically evaluating the ability of ultrasound in combination with air bubbles to evaluate neovascularisation in carotid artery plaques, the examination will be performed twice with an interval of 1/2 hour on the day before surgery, thus studying the reliability of the method.

The second goal of this study is to investigate whether MRI at 3.0 T with a custom-designed 3T carotid coil, using a recently developed pulse sequence, is able to accurately identify and quantify neovascularisation. And the third goal of this study is to make an intermodality comparison of CE-US and MRI regarding their ability to identify and quantify plaque neovascularisation.

DETAILED DESCRIPTION:
Atherosclerosis is a systemic disease of the large arteries and the leading cause of death in Western society. The development of atherosclerosis involves the accumulation of lipids, cells and extracellular matrix in the blood vessel wall. It is a progressive disease characterized by the formation of a fibrous cap by smooth muscle cell proliferation and migration, and the development of a necrotic/lipid core. This core develops due to the accumulation of lipids and apoptosis of lipid-loaded macrophages. In this process the intima, the innermost layer of the blood vessel, thickens. This will lead to narrowing of the lumen and obstruction of blood flow. The developed lesion of the vessel wall may become vulnerable to rupture of the fibrous cap. Cap rupture exposes the necrotic core to the blood leading to the formation of a thrombus. The thrombus may fully or partially obstruct the lumen and cause cardiovascular complications, such as myocardial infarction or stroke. Although atherosclerosis forms the origin of most cardiovascular diseases, at present much remains unknown of the atherogenic process. Therefore, it is essential that research is done to discover novel mechanisms of atherosclerotic development. Intimal neovascularisation has recently drawn much attention as a novel factor, likely contributing to atherosclerotic plaque growth and rupture. Neovascularisation occurs when the intima thickens and is associated with stenosis, plaque inflammation and hemorrhage. Because increased amount of neovascularisation may be associated with increased risk for stroke, it would be highly desirable to identify plaque neovascularisation by noninvasive imaging. At present, imaging of neovascular development in atherosclerotic lesions with conventional ultrasound is not feasible, since the vessel diameter is well below the resolution capacity of currently available ultrasound systems. Since almost a decennium, contrast-enhanced ultrasound (CE-US) with gaseous ultrasound contrast agents has been used for research purposes but is now also widely commercially available and registered for clinical use, which can be done safely. With the help of such a gaseous contrast medium containing air bubbles smaller than erythrocytes (microbubbles) it might be possible to depict neovascularisation in a carotid artery plaque, due to the strong signal that will be evoked even by a small number of air bubbles as compared to the signal from the surrounding tissue. So, the intensity increase of the ultrasound signal from the carotid artery plaque after administration of microbubbles might reflect the amount of neovascularisation. Until now, only case reports concerning this technique have been published, especially no comparison with histology has been performed. So, the first goal of this study is to investigate whether CE-US is able to accurately identify and quantify neovascularisation in carotid artery plaques. Since this is one of the first studies systematically evaluating the ability of ultrasound in combination with air bubbles to evaluate neovascularisation in carotid artery plaques, the examination will be performed twice with an interval of 1/2 hour on the day before surgery, thus studying the reliability of the method. Magnetic resonance imaging (MRI) is well suited for evaluating carotid plaques; it is widely available, provides excellent soft tissue contrast, multiplanar imaging capability, and is free of ionising radiation. Multisequence MRI has shown to be able to detect different carotid plaque components in vivo. However, only very little experience exists in identifying neovascularisation by MRI. Also, newer MRI systems (>1.5 T), newer coil systems, and better pulse sequences have recently become available. Therefore, the second goal of this study is to investigate whether MRI at 3.0 T with a custom-designed 3T carotid coil, using a recently developed pulse sequence, is able to accurately identify and quantify neovascularisation. Finally, the third goal of this study is to make an intermodality comparison of CE-US and MRI regarding their ability to identify and quantify plaque neovascularisation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a >70% carotid artery stenosis who are scheduled for carotid endarterectomy. Such subjects will be eligible if the subject's attending physician of the department of surgery concurs with this assessment.
* Age 18 years or older
* Informed consent by signing informed consent form regarding this study

Exclusion Criteria:

* Known hypersensitivity to sulphur hexafluoride or to any of the components of SonoVue.
* Acute coronary syndrome or clinically unstable ischaemic cardiac disease, including: evolving or ongoing myocardial infarction, typical angina at rest within last 7 days, significant worsening of cardiac symptoms within last 7 days, recent coronary artery intervention or other factors suggesting clinical instability (for example, recent deterioration of ECG, laboratory or clinical findings), acute cardiac failure, Class III/IV cardiac failure, or severe rhythm disorders.
* Right-to-left shunts, severe pulmonary hypertension (pulmonary artery pressure >90 mmHg), uncontrolled systemic hypertension, and adult respiratory distress syndrome.
* Pregnant and lactating women
* Documented allergy to contrast media or a renal clearance <30 ml/minute
* Standard contra-indications for MRI (ferromagnetic implants like pacemakers or other electronic implants, metallic eye fragments, vascular clips, claustrophobia, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Plaque neovascularization at contrast-enhanced ultrasound and MRI | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Werner H Mess, MD, PhD, Principal Investigator — Department of Clinical Neurophysiology, University Medical Center Maastricht
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands